CLINICAL TRIAL: NCT05290051
Title: Etude Prospective Comparative Des Performances de Détection Des Variations de Nombre et de Structure Des Chromosomes Par Les Techniques de Cartographie Moléculaire et de Séquençage de Grands Fragments
Brief Title: Prospective Study to Assess Medical Performance of Optical Mapping and Long Read Sequencing in Detecting Numerical and Structural Chromosome Abnormalities
Acronym: CHROMAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: CHU Rennes - Hopital Pontchaillou (Other); APHP (Other); CHU de Rouen - Accueil (Other); University Hospital, Strasbourg (Other); Université Montpellier (Other); University Hospital, Clermont-Ferrand (Other); CHU de Reims (Other); APHM (Unknown); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C21-35
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Infertility; Intellectual Disability; Malformation; Miscarriage
MeSH Terms: conditions — Infertility; Intellectual Disability; Congenital Abnormalities; Abortion, Spontaneous | interventions — Nanopores

STUDY DESIGN:
Intervention Model Description: Comparison of new diagnostic procedures with gold standard used in clinical setting
Masking Description: Gold standard analyses run as usual with results issued to patients Evaluated analyses run and analyzed blind to care provider and investigator Comparison of results between gold standard and tested analyses at the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients referred for cytogenetic analysis (Experimental): Analysis of patient DNA with Optical Genome Mapping (Bionano®) and long read Sequencing (Nanopore®) in search for chromosome abnormalities (aneuploidies and SV)
  Interventions: Genetic: Optical Genome Mapping (Bionano®); Genetic: Longread sequencing (Nanopore®)

INTERVENTIONS:
Genetic: Optical Genome Mapping (Bionano®) — Search for chromosome abnormalities through alteration of the optical map of the genome compared to reference genome using the Bionano® 's pipeline.
Genetic: Longread sequencing (Nanopore®) — Search for chromosome abnormalities from the sequencing data obtain from high molecular weight DNA molecules using dedicated analysis pipeline.

SUMMARY:
Chromosomal aberrations are major causes of developmental disorders (Intellectual disability (ID), multiple congenital anomalies (MCA), autism spectrum disorders (ASD)) as well as reproductive disorders (RD) in particular gametogenesis defects and recurrent miscarriages. Current first tier genetic investigations for chromosome analysis in clinical settings include karyotyping in case of RD (5 ~ 10% diagnosis rate) and chromosomal microarrays (CMA) in case of ID/MM (10 ~ 20% diagnosis rate). However, both assays show significant drawbacks, e.g. low resolution for karyotyping and inability to detect balanced structural rearrangement for CMA.

Optical genome mapping and long read genome sequencing are emerging technologies that offer new opportunities to overcome these limitations and allow for a higher resolution chromosome analysis.

This project aims at assessing the performance of optical mapping and long read whole genome sequencing compared to current gold standard cytogenetics methods in a prospective study. The investigator will evaluate their ability to become the all-in-one methodology for genomic analysis that could replace both karyotype and CMA and their added-value compared to these latter by uncovering new diagnoses.

DETAILED DESCRIPTION:
Chromosome aberrations are found in up to 1% of the general population. Structural aberrations, either balanced (3.6‰) or unbalanced (0.9‰), represent a third of them. Most (but not all) unbalanced anomalies are associated with a relevant phenotype, while most (but not all) balanced rearrangements have no consequence on the phenotype except possible reproductive disorders. Indeed, the prevalence of the latter among infertile individuals is ten times higher than in the fertile population. Moreover, 6% - 27% of apparently balanced rearrangements can lead to developmental disorders through various mechanisms.

First tier chromosome analysis methods, karyotype and chromosomal microarray analysis (CMA), are hampered either by a low resolution (karyotype) or by their inability to detect balanced rearrangements (CMA). However, karyotyping is still the gold standard analysis in case of reproductive disorders (RD) and recurrent miscarriages because of the high prevalence of aneuploidies (mainly sex chromosome aneuploidies, i.e. 45,X or 47,XXY) or balanced structural abnormalities.

According to a French national annual survey carried out by the Agence de la Biomedecine, the diagnostic yield is ~5%-10% for karyotyping in RD and ~15-20% for CMA in ID/MCA. Hence, many patients remain without a molecular diagnosis of their condition after these first tier studies. Whole exome sequencing and now whole genome sequencing have been shown to be able to rise the diagnostic yield to up to 50-60% in ID patients. However, current short read sequencing methods fall short to providing robust data for structural variation (SV) detection, because of the inability of bioinformatic tools to map correctly the sequences due to the high proportion of homologous sequences at SV breakpoints. New emerging methodologies based on long DNA fragments are now available and may provide a way to circumvent current limitations: long read sequencing (lrNGS) and optical genome mapping (OGM) :

OGM has been developed by Bionano Genomics and combines microfluidic and high-resolution microscopy to offer an imaging of long, high molecular weight, DNA molecules (up to more than 1Mb) labelled with specific sequence tags. From these images, a de novo assembly of any patient's genome can be performed and compared to a reference genome map to unravel all kind of structural rearrangements with a resolution that is 100 to 1000 times higher than with karyotyping. A second pipeline based on coverage in each region allows for the detection of large CNVs and aneuploidies.

lrNGS of long DNA fragments (several kb) reduces short read sequencing based assembly issues due to repetitive sequences, and allow for detection of all mutations, from SNVs to SVs and CNVs. Due to the large size of fragment inserts, less false positive are expected for SV calling than observed with short read or linked-read sequencing. Although bioinformatics pipelines are improving, prospective detection of large SV/SNV remains challenging, with a very high rate of false positives and false negatives. Furthermore, no study has been conducted to test prospectively the feasibility and medical efficiency of using long read sequencing as a first-tier all-in-one test for SV and CNV identification.

Primary Objective The main objective of this prospective study is to compare the diagnosis rate of OGM (Bionano®) and lrNGS (Nanopore®) to the one of standard-of-care technologies, e.g. karyotyping for patients presenting with reproductive disorders (primary amenorrhea, premature ovarian insufficiency, severe oligozoospermia, azoospermia) or CMA in case of developmental disorders (ID/MCA).

Secondary Objectives Refine the data on the incidence and type of chromosomal aberrations in the different clinical categories of patients Assess the limits of Bionano® and Nanopore® Assess the impact of enhanced detection of subchromosomal anomalies by Bionano® or Nanopore® on the medical care of the patient Compare the cost-effectiveness of both approaches

Study type This is a national multicentric prospective cohort study involving 14 French certified constitutional cytogenetic centers. The same patients will be offered genome wide analysis using standard techniques (Karyotyping or CMA according to the reason for referral) and two new genome wide analysis methods, OGM (Bionano®) and lrNGS (Nanopore®).

ELIGIBILITY:
Inclusion Criteria: patient requiring chromosome analysis either in case of infertility or in case of Intellectual deficiency/malformation

-

Exclusion Criteria: no exclusion criteria but we defined Non-inclusion criteria

* ID in a context of perinatal suffering (e.g. hypoxia during labor)
* Children born to non-native French-speaking parents in case of speech/language retardation
* Obstructive azoospermia
* Children under 5kg or whenever blood sampling cannot meet the required volume.
* Missing or wrong blood collection tube
* Insufficient blood volume
* Missing or incomplete consent to research (e.g. only one parental consent for a child)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of verified clinically significant chromosomal aberrations detected by Bionano® and Nanopore® compared to the percentage of those detected by karyotyping or CMA according to reason for referral. | Through study completion, an average of 1 year
  The significance of an aberration is assessed according to international guidelines, clinical history, as well as publications and public databases.

SECONDARY OUTCOMES:
Incidence and distribution of different kinds of chromosomal aberrations per category of referral. | Through study completion, an average of 1 year
  Two main referral indication: infertility or Intellectual deficiency/Malformation
Type of chromosome abnormalities that are overlooked by Bionano® and/or Nanopore® while detected by standard-of-care techniques | Through study completion, an average of 1 year
  Abnormalities detected with either karyotype or CMA and not by OGM (Optical Genome Mapping) or longread sequencing
Percentage of patients for which the detection of a chromosomal aberration by Bionano® or Nanopore® and not by karyotyping or CMA resulted in a change in the disease management | Through study completion, an average of 1 year
  Abnormalities detected by either OGM or lrNGS but not by gold standard techniques leading to a change in patient care (including genetic counselling).
Overall cost and benefit of each technique including delay to diagnosis and changes in the disease management | Through study completion, an average of 1 year
  Medico-economic evaluation of the new technologies compared to gold standard diagnostic tools.

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin APHP, Paris, France